CLINICAL TRIAL: NCT00140114
Title: Sublingual Versus Vaginal Misoprostol for Labor Induction at Term
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OGY.AN.02
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2008-08

CONDITIONS: Induction of Labor
Keywords: Vaginal, sublingual, misoprostol, cervical ripening
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): A: Vaginal misoprostol (cytotec)
  Interventions: Drug: Misoprostol (Cytotec®)
- B (Other): Sublingual misoprostol (Cytotec)
  Interventions: Drug: Misoprostol (Cytotec®)

INTERVENTIONS:
Drug: Misoprostol (Cytotec®) — 50 micrograms of sublingual or vaginal misoprostol every 4 hours for a maximum of 5 doses
  Other Names: Cytotec

SUMMARY:
Misoprostol (Cytotec®) is a synthetic prostaglandin E1 analog that has been marketed in the United States since 1988 as a gastric cytoprotective agent. In contradistinction to prostaglandin E2 preparations (dinoprostone, Prepidil, Cervidil), misoprostol is inexpensive and available in scored tablets that can be broken and inserted vaginally. Despite a focused campaign by the manufacturer to curtail its use in obstetric practice, misoprostol has, over the past several years, gained widespread acceptance as both a labor induction and a cervical ripening agent. Such off-label indication has been endorsed by the American College of Obstetricians and Gynecologists and other medical bodies. Recently, FDA approved a new label for the use of cytotec during pregnancy which removed pregnancy as a contraindication for its use. Vaginal administration seems to be more efficacious than when given orally, although there is the worry of uterine tachysystole and hyperstimulation with vaginal doses > 50-µg. The use of sublingual misoprostol for cervical ripening at term was recently investigated in two studies that compared it to the oral route, on the assumption that the sublingual route would have the higher efficacy of the vaginal route by avoiding the first pass effects of the gastrointestinal and hepatic systems, while having lower hyperstimulation rates by avoiding the direct effects on the cervix. In addition, the sublingual route would combine an easier administration with the added advantage of no restriction of mobility after administration. There has been no previous report in the literature comparing the use of misoprostol given sublingually to that given vaginally for the induction of labor at term. Our aim is to compare efficacy, safety and patient satisfaction with misoprostol given vaginally (the current standard) to that given sublingually.

DETAILED DESCRIPTION:
Misoprostol, a synthetic prostaglandin E1 analog, has been given both orally and vaginally for induction of labor in the third trimester.1 Vaginal misoprostol has been shown to be more efficacious than oral misoprostol in equivalent doses,2 although there is the worry of uterine tachysystole and hyperstimulation with vaginal doses of 50 µg or higher.2-4 The higher efficacy after vaginal administration may be explained by the pharmacokinetics of the drug. Zeiman et al5 showed that the systemic bioavailability of vaginally administered misoprostol is 3 times higher than that after oral administration. Plasma concentrations of its metabolite, misoprostol acid, peak one to two hours after vaginal application as compared with the peak seen 30 minutes following oral administration, and although peak levels are lower with the vaginal route, they are sustained longer and overall exposure to the drug is increased, perhaps because of the presystemic gastrointestinal or hepatic metabolism that occurs with the oral route. An additional explanation for the higher efficacy could be that there is a direct effect on the cervix that initiates the physiologic events that lead to increased uterine contractility.6 However, there seems to be a trend toward patient preference for the oral route. The sublingual route of administration has not been reported in the literature prior to 2001. Since then and partly because of issues relating to patient preference, investigators started studying the sublingual route of administration of misoprostol. In theory, the sublingual route could mimic vaginal administration pharmacokinetically, although there have been no such reported studies on this route of administration.

It is speculated that sublingual misoprostol could combine the higher efficacy of the vaginal route by avoiding gastrointestinal and hepatic metabolism, but it could have a more restrained effect on uterine contractility by avoiding direct effects on both the uterus and cervix. Therefore, in theory, the sublingual route may have lower hyperstimulation rates and would have the advantage of a less invasive administration and lack of restriction of mobility.

Although many studies have been published on the use of sublingual misoprostol for medical abortion in the first and second trimesters, 7-11, only two studies (by the same group) have compared sublingual to oral misoprostol, in different doses.12,13 The 50-µg dose was chosen because it is the dose most commonly used orally and vaginally in various studies reported in the literature.3,14 To the best of our knowledge, no study comparing sublingual to vaginal misoprostol for labor induction at term has been previously published in the literature. Therefore, this study, when completed will provide evidence on the relative effect and safety profile of different routes of administration of misoprostol for labor induction.

The aim of our study is to compare the efficacy of a 50-µg sublingual dose of misoprostol administered at 4-hour intervals with an equivalent dose regimen administered vaginally in women admitted for induction of labor for a medical or obstetric indication at term. In addition, we want to assess the safety profile and patient acceptability of the 2 modes of administration.

The study hypothesis is that the sublingual route of administration of misoprostol is as effective as the vaginal route for induction of labor at term and is more acceptable to patients as compared to vaginal misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* Live singleton pregnancy at a gestational age of 36 wks or more with a medical or obstetric indication for induction
* Both nulliparous and multiparous women
* A cephalic presentation
* An unfavorable cervix (Bishop's score less than 8)
* A reassuring fetal heart tracing.

Exclusion Criteria:

* Rupture of membranes
* Multiple gestation
* Malpresentation (presentation other than cephalic)
* Previous cesarean delivery
* Known contraindications to the use of prostaglandins (e.g. asthma)
* Grandmultiparity (more than 5)
* Significant fetal or maternal concerns that made induction necessary under continuous monitoring (e.g. severe IUGR, severe preeclampsia)

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2004-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The proportion of women satisfied with the route of administration of misoprostol. | 48 hours of enrollment

SECONDARY OUTCOMES:
The interval of induction to delivery | Within 24 hours of induction
Number of doses of misoprostol given | Within 24 hours of induction
Number of unsuccessful inductions | Within 24 hours of induction
Number of cesarean deliveries for fetal concerns | Within 24 hours of randomization
The incidence of tachysystole | within 24 hours of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Anwar H Nassar, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon